CLINICAL TRIAL: NCT00391521
Title: A Phase I Multicenter, Open-Label, Dose Escalation Trial of AS703569 Given Orally to Subjects With Solid Tumours
Brief Title: AS703569 Phase I in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26865
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Solid Tumors
Keywords: Oncology. All solid Tumour disease.
MeSH Terms: interventions — MSC1992371A

ARMS (3):
- 1 (Active Comparator): Regimen 1
  Interventions: Drug: AS703569
- 2 (Active Comparator): Regimen 2
  Interventions: Drug: AS703569
- 3 (Active Comparator): Regimen 3
  Interventions: Drug: AS703569

INTERVENTIONS:
Drug: AS703569 — Regimen 1: 3 mg/m2 /day given orally on Days 1 and 8 during a 21-day cycle
  Other Names: MSC1992371A; Aurora kinase inhibitor
  Arms: 1
Drug: AS703569 — Regimen 2: 2 mg/m2/day given orally on Days 1, 2, and 3 of a 21-day cycle
  Other Names: MSC1992371A; Aurora kinase inhibitor
  Arms: 2
Drug: AS703569 — Regimen 3: 10 mg/m2/day given orally on Days 1, 2, 3 and Days 8, 9, 10 of a 21-day cycle
  Other Names: MSC1992371A; Aurora kinase inhibitor
  Arms: 3

SUMMARY:
This is a Phase I trial. Some specific protocol information is proprietary and is not publicly available at this time. Full information will be provided to trial participants.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed locally advanced or metastatic solid tumour that is either refractory after standard of care therapy for the disease or for which standard of care therapy is not reliably effective or has a cancer for which no standard therapy exists
2. Age greater than or equal to 18 years
3. Has read and understands the informed consent form and is willing and able to give informed consent, and subject authorization under Health Insurance Portability and Accountability Act (HIPAA). Fully understands requirements of the study and willing to comply with all study visits and assessments
4. Subjects and their partners must be willing to avoid pregnancy during the study and until 1 month after the last study drug administration. Males with female partners of childbearing potential and female subjects of childbearing potential must therefore be willing to use adequate contraception such as, intra uterine device, diaphragm, or condom, for the duration of the study. For the purposes of this study, childbearing potential is defined as: "All female subjects unless they are post- menopausal for at least two years, are surgically sterile or sexually inactive"
5. Negative serum pregnancy test at the screening visit for women of childbearing potential

Exclusion Criteria:

1. Bone marrow impairment as evidenced by Hb < 9.0 g/dl, ANC < 1.5x 109/L, platelets < 75 x 109/L. Subjects may be transfused.
2. Renal impairment as evidenced by serum creatinine > 1.5 x ULN (upper limit of normal), and/or calculated creatinine clearance < 60 ml/min
3. Liver function abnormality as defined by total bilirubin > 1.5 ULN, or AST or ALT > 2.5x ULN at screening; for subjects with liver involvement AST or ALT > 5x ULN at screening
4. INR (blood coagulation) > 1.5 x ULN for subjects not on therapeutic doses of coumadin
5. History of CNS metastases, unless subject has been previously treated for CNS metastases, is stable by CT scan without evidence of cerebral edema, and has no requirements for corticosteroids or anticonvulsants
6. History of difficulty swallowing, malabsorption or other chronic gastro- intestinal disease or conditions that may hamper compliance and/or absorption of the tested product
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) > 2
8. Known HIV, hepatitis C, or hepatitis B positivity
9. Has received chemotherapy, immunotherapy, hormonal therapy, biologic therapy, or any other anticancer therapy or surgical intervention within 28 Days of Day 1 of study drug treatment (6 weeks for nitrosureas or mitomycin C), and must have fully recovered
10. Has received extensive prior radiotherapy on more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation
11. Has received any investigational agent within 28 days of Day 1
12. Has history of any other significant medical disease or intervention including major gastric or small bowel surgery or has a psychiatric condition that might impair the subjects well-being or preclude full participation in the study
13. Is a pregnant or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects experiencing: at least a Dose-Limiting Toxicity (DLT) in each cohort during the first cycle. | Undefined

SECONDARY OUTCOMES:
Plasma and urine PK parameters of AS703569, genetic markers and potential markers of clinical and biological response. | Undefined
Number and proportion of subjects with Progressive Disease as assessed at the end of every other cycle. | Undefined

CONTACTS AND LOCATIONS:
Overall Officials: Narmyn Rejeb, MD, Study Director — Merck Serono S.A., Geneva
Locations (1):
- EMD Serono Medical Information Office, Rockland, Massachusetts, United States

REFERENCES:
- [Result] Mita M, Gordon M, Rejeb N, Gianella-Borradori A, Jego V, Mita A, Sarantopoulos J, Sankhala K, Mendelson D. A phase l study of three different dosing schedules of the oral aurora kinase inhibitor MSC1992371A in patients with solid tumors. Target Oncol. 2014 Sep;9(3):215-24. doi: 10.1007/s11523-013-0288-3. Epub 2013 Jul 6. PMID 23832397